CLINICAL TRIAL: NCT00270192
Title: The Effects Of Antenatal Breast Preparation On The Successful Initiation And Continuation Of Breastfeeding In Singaporean Mothers
Brief Title: Antenatal Educational Intervention for Improvement of Breastfeeding
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Educational/Counseling/Training
Other Study IDs: NHG RPR 01101
Record Dates: First submitted 2005-12-23; First posted 2005-12-26 (Estimated); Last update posted 2006-10-24 (Estimated); Status verified 2005-12

CONDITIONS: Breastfeeding
Keywords: Breastfeeding; exclusive; education; counseling
MeSH Terms: conditions — Breast Feeding

INTERVENTIONS:
Behavioral: individual lactation counseling and educational material
Behavioral: educational material alone
Behavioral: routine antenatal care without educational intervention

SUMMARY:
This randomized controlled trial addresses the impact of simple antenatal breastfeeding educational interventions on breastfeeding rates and practice in a tertiary hospital setting.

Hypothesis: A single antenatal encounter, which includes breastfeeding educational material and individual instruction with a lactation counselor, can improve the initiation, duration and exclusivity of breastfeeding compared to routine antenatal care or the use of educational material alone

DETAILED DESCRIPTION:
Breastfeeding rates in many developed countries, particularly in terms of exclusive and predominant breastfeeding, often fall short of the recommended practice advised by the World Health Organization and the American Academy of Pediatrics. Despite increasing awareness of the many advantages of breastfeeding the challenge remains to implement programs that can effectively improve short and long-term breastfeeding rates.

The Singapore National Breastfeeding Survey 2001 (Foo et al, 2005) demonstrated an encouraging breastfeeding initiation rate of 94.5%. However only 21.1% continued to breastfeed at 6 months with fewer than 5% breastfeeding exclusively.

The formal preparation of expectant mothers for breastfeeding is not part of routine antenatal care in many practices. We feel that it may prove beneficial especially in an environment with a low prevalence of breastfeeding. The aim of this trial is to demonstrate the impact of single-encounter antenatal education combining educational material with individual instruction, on breastfeeding initiation and duration and on infant feeding practice, compared with routine antenatal care and educational material alone in a tertiary hospital setting.

401 women are randomized into 3 predetermined groups and are exposed to specific antenatal education materials targeting breastfeeding techniques; the control group receives routine antenatal care. Data regarding breastfeeding rate, quality and duration is collected over a 1 year period.

Comparisons: breastfeeding initiation rate, duration and type among women receiving lactation counseling with educational material, educational material without individual counseling, and routine antenatal care without educational intervention

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy
* gestation of at least 36 weeks at recruitment
* no uterine scar
* the absence of any obstetric complication that would contraindicate vaginal delivery.

Exclusion Criteria:

* refusal to participate in trial
* contraindications to labour, vaginal delivery, breastfeeding

Ages: 21 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 450
Dates: Start 2002-05; Study Completion 2004-12

PRIMARY OUTCOMES:
Comparison of exclusive or predominant breastfeeding rates in intervention groups versus controls

SECONDARY OUTCOMES:
Breastfeeding initiation, defined as any breastfeeding type within the first 2 weeks of delivery

CONTACTS AND LOCATIONS:
Overall Officials: Yah Shih Chan, MHSc, Principal Investigator — National University Hospital, Singapore; Citra N Mattar, MRANZCOG, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Background] Foo LL, Quek SJ, Ng SA, Lim MT, Deurenberg-Yap M. Breastfeeding prevalence and practices among Singaporean Chinese, Malay and Indian mothers. Health Promot Int. 2005 Sep;20(3):229-37. doi: 10.1093/heapro/dai002. Epub 2005 Apr 6. PMID 15814526